CLINICAL TRIAL: NCT06826456
Title: Effect of Er,Cr:YSGG Sub-Ablative Laser Irradiation on Fissure Caries Prevention in Permanent Molars
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Hussein Ezz, Assistant Lecturer, Pediatric dentistry department, Faculty of dentistry, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10556-0008839
Record Dates: First submitted 2025-01-30; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Caries,Dental
Keywords: Er,Cr:YSGG; laser; DIAGNOdentTM; acid resistance
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Laser irradiation (Experimental): First permanent molars subjected to sub-ablative Er,Cr:YSGG laser
  Interventions: Procedure: sub-ablative Er,Cr:YSGG laser
- Fluoride Varnish (Active Comparator): First permanent molars subjected to fluoride varnish application
  Interventions: Procedure: Fluoride varnish application

INTERVENTIONS:
Procedure: sub-ablative Er,Cr:YSGG laser — The irradiations will be done with an Er,Cr:YSGG laser device Er,Cr:YSGG Laser (Waterlase iPlus 2011,Biolase,Germany). This equipment emits photons at a wavelength of 2.78 µm. The repetition rate will be fixed at 20 Hz. The pulse duration will be fixed on 140 µs. The beam diameter at the focal area for the handpiece will be 600 µm. The tip will be positioned 1.0 mm from the enamel surface (focused mode). The handpiece will be positioned perpendicularly to the enamel. Power =0.25 Watt; energy density per pulse will be 62.5 J/cm2, Time = 20 seconds; Frequency = 20 Hz; without air/water. To ensure that each spot of a fissure was irradiated, each fissure will be irradiated for 2 min with overlapping irradiation
  Arms: Laser irradiation
Procedure: Fluoride varnish application — The first permanent molar assigned for control group will receive fluoride varnish applications. Fluoride varnish will be applied to all teeth in the oral cavity, including the laser-treated as well as the control tooth at baseline and the 6-month recall.
  Parents and children will be given age-appropriate oral hygiene instructions including proper teeth brushing with a 1100-ppm fluoride-containing dentifrice for at least 2 min twice daily especially before bedtime, as well as flossing if indicated.
  Arms: Fluoride Varnish

SUMMARY:
Background: Subjecting human dental enamel to sub-ablative laser has been suggested as a novel way of caries prevention. However, further studies are needed to establish its use as a routine clinical procedure for caries prevention.

The aim of this study: This study aims to evaluate the effect of Er,Cr:YSGG subablative laser irradiation on caries resistance of occlusal fissures of permanent molars.

Materials and methods: In-vivo study, a split mouth randomized controlled trial with sixty patients having two fully erupted bilateral first permanent molars (ICDAS-II score 0,1 or 2). The pits and fissures will be subjected to sub-ablative power of Er,Cr:YSGG Laser (Group 1, n=90) and will be compared with fluoride varnish application on the first permanent molars in the same arch(Group 2,n=90). DIAGNOdentTM readings and changes in ICDAS-II score will be assessed at base line and at 3,6,9 and 12 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Participants of age 6-12 years old
* Patients ranking definitely positive or positive on Frankl behavior rating scale
* Having at least two bilateral fully erupted first permanent molars with untreated non-cavitated occlusal surfaces with deep grooves, the included teeth will have International Detection and Assessment System (ICDAS-II)/ severity scores 0, 1 or 2
* Initial DIAGNOdent Score not exceeding value of 25 indicating only enamel involvement
* Patients whom their parents are willing to comply with all study procedures and protocols and will be given an informed consent to participate

Exclusion Criteria:

* Patients with any known medical history of systemic diseases
* Patients having first permanent molar with hypoplastic or hypocalcified enamel
* Patients using medications that may affect the oral flora or salivary flow
* Patients treated with in-office fluoride treatment within the last 3 months prior to being enrolled in the study.
* Patients showing evidence of poor oral hygiene according to Silness and Löe plaque index

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Diagnodent scoring | day 0, 3 months, 6 months, 12 months
  evaluate the dental caries activity of fissures by comparing changes in DIAGNOdent readings. Laser induced fluorescence (DIAGNOdentTM) will be used to quantitatively determine lesion demineralization which is displayed as numerical values ranging from 0 to 99. A decrease in the signal indicates regression of the carious lesion, whereas an increase indicates progression. The DIAGNOdent tip will be then placed on the measurement site, and slightly tilted circular movements will be performed along the entire fissure pattern. The patient will be included in the study if the DIAGNOdent readings of both bilateral first permanent molar do not exceed 25.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided